CLINICAL TRIAL: NCT01523184
Title: A Phase II, Single-Center, Randomized, Parallel Group, Multiple Administration, Double-Blind, Placebo-Controlled Study to Evaluate the Pharmacodynamics of YKP10811 in Patients With Chronic or Functional Constipation
Brief Title: A Phase 2 Study to Evaluate Pharmacodynamics of YKP10811 in Patients With Chronic or Functional Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YKP10811C003
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Constipation; Functional Constipation
Keywords: Chronic constipation (CC); Functional Constipation (FC); Gastric Emptying; Colon Transit; multiple doses of YKP10811; gastrointestinal transit; colonic transit

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo Capsule (Placebo Comparator): Placebo Capsules
  Interventions: Drug: Placebo Capsule
- YKP10811 Drug Product Capsule, 10 mg (Active Comparator)
  Interventions: Drug: YKP10811 Drug Product Capsule
- YKP10811 Drug Product Capsule, 20 mg (Active Comparator)
  Interventions: Drug: YKP10811 Drug Product Capsule
- YKP10811 Drug Product Capsule, 30 mg (Active Comparator)
  Interventions: Drug: YKP10811 Drug Product Capsule

INTERVENTIONS:
Drug: Placebo Capsule — This is the placebo capsule
  Arms: Placebo Capsule
Drug: YKP10811 Drug Product Capsule — The drug product, YKP10811, 10 mg under investigation
  Arms: YKP10811 Drug Product Capsule, 10 mg
Drug: YKP10811 Drug Product Capsule — The drug product, YKP10811, 20 mg under investigation
  Arms: YKP10811 Drug Product Capsule, 20 mg
Drug: YKP10811 Drug Product Capsule — The drug product, YKP10811, 30 mg under investigation
  Arms: YKP10811 Drug Product Capsule, 30 mg

SUMMARY:
This will be a single-center, randomized, parallel group, multiple dose administration, double-blind, placebo-controlled study to evaluate the effects of YKP10811 on gastric, small bowel, and colonic transit in patients with Chronic Constipation or Functional Constipation. Four groups including a placebo group will be enrolled and will receive multiple oral doses of YKP10811 or matching placebo.

DETAILED DESCRIPTION:
If the participant fulfills the initial eligibility criteria, the patient will be randomized to 1 of the active treatment groups or placebo. During the treatment period, patients will receive study medication once daily for 8 days. Patients will undergo scintigraphic assessment of gastric, small bowel and colonic transit of solids over the 48-hour period.

Patients will be males or females, 18 through 65 years of age with a body mass index (BMI) of 19 through 40 kg/m2, with Chronic Constipation or Functional Constipation and no evidence of evacuation disorder as assessed by the Investigator and meet all the inclusion criteria and none of the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smokers (refrained from any tobacco or nicotine usage, including smokeless tobacco, nicotine patches, etc.) for at least 6 months prior to Day 1 of the study
2. Body Mass Index of 19 through 40 kg/m2
3. Participants must be willing to follow dietary restrictions
4. Females of childbearing potential (ie, not menopausal, no hysterectomy, no bilateral oophorectomy) must complete a negative pregnancy test (urine) prior to receiving any radioisotopes
5. No evidence of pelvic floor dysfunction
6. If clinically indicated, absence of an evacuation disorder should be confirmed within 30 days prior to the first dose of study medication
7. At Screening, patients must meet ROME III Criteria for FC, which assumes an absence of a structural or biochemical explanation
8. The patient's screening (baseline) colonic transit test must show a GC ≤ 2.4 at 24 hours; and
9. Baseline EKG shows QTc interval ≤ 450mSec

Exclusion Criteria:

1. History of clinically-significant manifestations or current abnormality of any organ system
2. History of inflammatory bowel disease
3. Any history of GI surgery within 6 months prior to the first dose of study medication
4. History of clinically-significant prolonged diarrhea, in the absence of a laxative
5. Patients who have started a special dietary habit and/or an intense physical workout program within 4 weeks prior to the first dose of study medication
6. Any clinically-significant surgical procedure within 30 days prior to the first dose of study medication
7. History of alcoholism or drug addiction within 12 months prior to the first dose of study medication
8. Any patient who has had an acute illness within 5 days prior to the first dose of study medication, eg, flu syndrome, GI virus, indigestion
9. Patients who are breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Colonic Geometric Center (GC) at 24 hours | 48 hours
  The colonic GC at 24 hours is the measurement of the move of the food within the GI track.

SECONDARY OUTCOMES:
Gastric emptying half time | 4 hours
  The gastric emptying half time is the time to empty the half of the ingested solid food in the stomach.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Shin A, Acosta A, Camilleri M, Boldingh A, Burton D, Ryks M, Rhoten D, Zinsmeister AR. A randomized trial of 5-hydroxytryptamine4-receptor agonist, YKP10811, on colonic transit and bowel function in functional constipation. Clin Gastroenterol Hepatol. 2015 Apr;13(4):701-8.e1. doi: 10.1016/j.cgh.2014.08.012. Epub 2014 Aug 19. PMID 25148765